CLINICAL TRIAL: NCT07054307
Title: MRG003 Plus HX008 as First-Line Treatment for EGFR-Positive Locally Advanced or Metastatic Penile Squamous Cell Carcinoma: A Prospective, Single-Arm, Phase I Clinical Trial
Brief Title: MRG003 Plus HX008 as First-Line Treatment for EGFR-Positive Locally Advanced or Metastatic Penile Squamous Cell Carcinoma
Acronym: MH-Penile-001
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiyan Liu (Other)
Collaborators: West China Hospital (Other); Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jiyan Liu, Deputy Director of the Department of Biotherapy, West China Hospital, Sichuan University, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MH-Penile-001; 274863 (Other: Chinese Clinical Trial Registry)
Record Dates: First submitted 2025-05-30; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Penile Cancer
Keywords: penile cancer; ADC; PD-1
MeSH Terms: conditions — Penile Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRG003 + HX008 arm (Experimental): MRG003 and HX008 will be administrated together.
  Interventions: Drug: MRG003; Drug: HX008

INTERVENTIONS:
Drug: MRG003 — MRG003 (2.3 mg/kg, IV, Q3W). Treatment continues until disease progression, intolerable toxicity, withdrawal, death, or sponsor termination.
Drug: HX008 — HX008 (200 mg, IV, Q3W). Treatment continues until disease progression, intolerable toxicity, withdrawal, death, or sponsor termination.

SUMMARY:
Penile squamous cell carcinoma (PSCC) is a rare malignancy, with stage IV patients exhibiting a 2-year overall survival (OS) rate of 21% and a 5-year survival rate of 0%. Both the National Comprehensive Cancer Network (NCCN) and European Association of Urology (EAU) guidelines recommend chemotherapy as the first-line treatment. However, the efficacy of chemotherapeutic agents in PSCC remains suboptimal, and options after chemotherapy failure are extremely limited. In recent years, targeted therapy and immunotherapy have demonstrated potential in treating this disease. Combination therapies based on chemotherapy, particularly chemoimmunotherapy combined with targeted therapy, have shown promising antitumor effects. Nevertheless, these regimens are associated with significant adverse effects and impose high physical demands on patients.

Therefore, this study aims to explore a "highly effective and low-toxicity" first-line treatment regimen for advanced PSCC patients. The objective is to evaluate the combined therapeutic efficacy of an epidermal growth factor receptor (EGFR)-targeted antibody-drug conjugate (MRG003) and an immune checkpoint inhibitor (HX008) through a single-arm, phase I, prospective clinical trial.

DETAILED DESCRIPTION:
Penile squamous cell carcinoma (PSCC) is a superficial tumor that could theoretically be detected early. However, due to social stigma and privacy concerns, patients often delay seeking medical attention until the disease reaches an advanced stage. For advanced PSCC, systemic therapy plays a crucial role in disease management. Currently, there is limited literature on palliative chemotherapy for advanced or recurrent cases, and prospective controlled studies are lacking.

Both the National Comprehensive Cancer Network (NCCN) and the European Association of Urology (EAU) guidelines recommend chemotherapy as the first-line treatment. However, chemotherapeutic agents show limited efficacy in penile squamous cell carcinoma, with single-agent response rates (e.g., bleomycin, methotrexate, 5-FU, cisplatin) below 20%. Treatment options after chemotherapy failure are also scarce. Combination chemotherapy regimens, such as TIP (paclitaxel, ifosfamide, cisplatin) or PF (cisplatin + 5-FU), demonstrate higher response rates (30-50%).

Based on our preclinical research and clinical experience, the investigators believe that investigating the efficacy and safety of combining EGFR-targeted therapy, immunotherapy, and chemotherapy in PSCC is warranted. This study aims to explore a novel and effective treatment option for EGFR-positive locally advanced or metastatic PSCC patients by combining an EGFR-targeted antibody-drug conjugate (MRG003) with a PD-1 inhibitor (HX008).

MRG003 is an EGFR-targeted ADC composed of three key components: Anti-EGFR monoclonal antibody (JMT101), Potent cytotoxic payload (monomethyl auristatin E, MMAE), and Cleavable linker (valine-citruline, vc linker). MRG003 is synthesized by conjugating chemically synthesized vc-MMAE with CHO cell-expressed JMT101.

HX008 is a novel neutralizing and blocking monoclonal antibody targeting human programmed death-1 (PD-1) independently developed by Hanchong Biotechnology. As a human immunoglobulin G4/kappa (IgG4/κ) subtype antibody, it exhibits high binding affinity to PD-1 and selectively blocks the interaction between PD-1 and its ligands programmed death-ligand 1 (PD-L1) and programmed death-ligand 2 (PD-L2), thereby activating T lymphocytes, enhancing lymphocyte proliferation, and promoting cytokine secretion, particularly interferon-gamma (IFN-γ). The primary pharmacodynamic studies of HX008 included in vitro PD-1 binding affinity assessment, cross-species binding specificity analysis, blockade of PD-1/PD-L1 and PD-1/PD-L2 interactions, T cell activation evaluation, as well as in vivo antitumor activity testing in both HCC827 human non-small cell lung cancer (NSCLC) xenograft models and PD-1 humanized genetically engineered mouse (HuGEMM) MC38 syngeneic colon tumor models. HX008 received clinical trial approval (No. 2017L04642) from China's National Medical Products Administration (NMPA) on August 28, 2017, and has since been undergoing multiple clinical trials in China for the treatment of various malignant tumors.

Clinical studies have demonstrated that the combination therapy of Adcetris® (Brentuximab Vedotin) and Nivolumab in a phase I/II clinical trial for relapsed or refractory Hodgkin lymphoma showed superior efficacy. Among 62 patients who received four cycles of combination treatment, 61% achieved complete response (CR), significantly higher than the CR rates of 34% and 9% observed with Adcetris® and Nivolumab monotherapies, respectively, indicating enhanced therapeutic benefits from the combination. When administered at their respective recommended phase II doses (RP2D) (BV 1.8 mg/kg, Nivo 3 mg/kg, every 3 weeks), the combination was well-tolerated, with a safety profile consistent with those of the individual agents. Additionally, increased levels of pro-inflammatory cytokines and chemokines were observed during combination therapy, suggesting synergistic effects between ADC and immunotherapy.

Similarly, preliminary results from a phase I clinical trial (NCT03288545) evaluating Padcev® (Enfortumab Vedotin) plus Pembrolizumab as first-line treatment for locally advanced or metastatic urothelial carcinoma demonstrated a significantly higher objective response rate (ORR) with the combination (71%) compared to Padcev® (44%) or Pembrolizumab (21%) monotherapies. At their respective RP2D doses (EV 1.25 mg/kg, Pembro 200 mg, every 3 weeks), the combination exhibited favorable tolerability, with a safety profile similar to that of each drug alone. These preclinical and clinical findings strongly support the synergistic antitumor effects of combining immune checkpoint inhibitors with ADCs, providing robust evidence for the potential of PD-1/PD-L1 immunotherapies in combination with ADC-based treatments.

This trial will evaluate the efficacy and safety of MRG003 (recombinant humanized anti-EGFR mAb-MMAE conjugate) combined with HX008 (recombinant humanized anti-PD-1 mAb) as first-line therapy in EGFR-expressing locally advanced or metastatic PSCC patients. MRG003 (2.3 mg/kg, IV, Q3W) and HX008 (200 mg, IV, Q3W) will be administrated on enrolled patients. Treatment continues until disease progression, intolerable toxicity, withdrawal, death, or sponsor termination. After treatment completion, all patients will undergo survival follow-up every 3 months until death, loss to follow-up, consent withdrawal, or study termination by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed unresectable, locally advanced, or metastatic penile squamous cell carcinoma.
2. EGFR expression (defined as IHC 1+, 2+, or 3+) confirmed by the institutional pathology department using primary or metastatic tumor tissue samples.
3. No prior systemic therapy for advanced disease.
4. Male, aged ≥18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 with a life expectancy ≥3 months.
6. At least one measurable lesion per RECIST 1.1 criteria.
7. Adequate organ function (based on institutional laboratory reference ranges):

   Left ventricular ejection fraction (LVEF) ≥50%.

   Hematology:

   Hemoglobin (HGB) ≥90 g/L, White blood cell count (WBC) ≥3.0×10⁹/L, Absolute neutrophil count (ANC) ≥1.5×10⁹/L, Platelet count (PLT) ≥80×10⁹/L.

   Biochemistry:

   Total bilirubin (TBIL) ≤1.5× upper limit of normal (ULN), AST/ALT ≤2.5×ULN (≤5×ULN if liver metastases present), Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (CrCl) ≥50 mL/min.
8. Willing to provide written informed consent, with full understanding of the study requirements and commitment to comply with trial procedures and follow-up visits.

Exclusion Criteria:

1. Patients who have received prior systemic therapy before enrollment.
2. History of other malignancies, except for cured carcinoma in situ of the cervix, basal cell carcinoma of the skin, or other malignancies that have been disease-free for at least 5 years.
3. Presence of central nervous system metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may be eligible if they have been stable for at least 6 months, show no disease progression on imaging within 4 weeks before treatment, have no neurological symptoms, demonstrate no evidence of new or enlarging brain metastases, and have discontinued radiation, surgery, or steroid therapy for brain metastases at least 28 days prior to the first dose. Carcinomatous meningitis is excluded regardless of clinical stability.
4. Severe or uncontrolled concurrent diseases, including uncontrolled infections, active tuberculosis, uncontrolled diabetes, cardiovascular diseases (such as NYHA Class III or IV heart failure, second-degree or higher heart block, myocardial infarction within the past 12 months, unstable arrhythmia or angina, or cerebral infarction within the past 6 months), pulmonary diseases (such as interstitial lung disease, chronic obstructive pulmonary disease, or a history of symptomatic bronchospasm), deep vein thrombosis or pulmonary embolism within the past 12 months, or decompensated cirrhosis.
5. Active autoimmune disease requiring systemic treatment (e.g., disease-modifying drugs, corticosteroids, or immunosuppressants) within the past 2 years. Replacement therapies (e.g., thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency) are permitted.
6. Positive serological virology test results, including HIV positivity, HBsAg positivity with detectable HBV DNA (≥2000 copies/mL), or HCV antibody positivity (eligible only if HCV RNA PCR-negative).
7. Major surgery within 4 weeks before enrollment, or prior allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
8. Administration of or plans to receive anti-cancer vaccines within 4 weeks before enrollment or during the study.
9. Clinically significant pleural effusion or ascites, as determined by the investigator to be unsuitable for enrollment.
10. Any other condition considered by the investigator to make the patient ineligible for the clinical study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biological males (assigned male at birth) are eligible due to penile-specific endpoints.
Enrollment: 10 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 weeks
  CT scans

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 12 weeks
  CT scans and follow-up by phone
Disease control rate (DCR) | 12 weeks
  CT scans
Duration of response (DoR) | 12 weeks
  CT scans and follow-up by phone
Overall survival (OS) | 12 weeks
  Follow-up by phone

IPD SHARING:
Plan to Share IPD: No